CLINICAL TRIAL: NCT01681238
Title: A Randomized Study of Goal-directed Therapy in the Elderly High-risk Patients Undergoing Total Hip Replacement
Brief Title: Goal-directed Therapy in High-risk Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, Professor, Vice Chair, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZZD-025
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Perioperative/Postoperative Complications; Hypovolemia; Hypoxia
Keywords: perioperative fluid optimization; goal-directed therapy; elderly; high-risk surgery
MeSH Terms: conditions — Postoperative Complications; Hypovolemia; Hypoxia | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Protocol group 1 (Other): Using standard hemodynamic therapy
  Interventions: Procedure: Protocol group 1
- Protocol group 2 (Experimental): Using goal-directed therapy
  Interventions: Procedure: Protocol group 2

INTERVENTIONS:
Procedure: Protocol group 2 — ensure SpO2≥ 92%, MAP 65-100 mmHg, HR <100 bpm, Hb> 8mg/dL and temperature ≥ 36℃, the patients were then administrated a 200 ml colloid as a fluid challenge. The fluid challenge repeat until the SV failed to increase by a factor of 10%. If at this stage the DO2I can not be greater than 600 mL/m2, then dobutamine will be started at a dose of 2.5 μg/kg/min and increased by the same increment every 20 minutes until the described target is reached or until a maximal dose of 20 μg/kg/min is given. Dobutamine is decreased in dose or discontinued if the heart rate is above 120 beats per minute or shows signs of cardiac ischemia. Blood transfusions will be used to maintain a hemoglobin concentration over 8mg/dL
  Other Names: goal-directed therapy
  Arms: Protocol group 2
Procedure: Protocol group 1 — The goal of this protocol is to ensure MAP> 65 mmHg, CVP 8-12 cmH2O. If meet the above requirements, do nothing, re-evaluate after 5min. If CVP <8 cmH2O, the patient will receive an additional 200ml colloid .If MAP beyond the scope of 65-100 mmHg, vasoactive agents will be administrated until achieve the goal. If 25mL/kg colloid given before goal is achieved, fluid challenges will then be performed with 200mL boluses of Ringer's lactate solution. Blood transfusions will be used to maintain a hemoglobin concentration over 8mg/dL
  Other Names: conventional fluid management
  Arms: Protocol group 1

SUMMARY:
There is growing evidence that the risk of postoperative complications can be decreased by optimizing the amount and type of infusion fluids given during surgery, steered by goal-directed therapy based on flow-related hemodynamic parameters, particularly in high-risk patients. This study is undertaken subsequently to test the hypothesis that the intraoperative goal-directed strategy based on FloTrac/Vigileo, a minimally invasive monitor, can partially prevented postoperative complications and shorten hospital stay in the elderly high-risk patients undergoing total hip replacement with continuous spinal anaesthesia .

DETAILED DESCRIPTION:
After sedated with IV 0.02 mg/kg midazolam, all patients will receive arterial, central venous, and L3-4 intrathecal catheterizations. A T12 sensory level block was attained with ropivacaine through the intrathecal catheter. Besides currently recommended monitoring during the intraoperative period, arterial blood pressure, stroke volume (Edwards Lifesciences, Irvine, Calif.), and central venous oxygen saturation (Edwards Lifesciences) will be measured and recorded. All Patients will receive intranasal oxygen 2 mL/min and be kept normothermic (body temperature > 36°C). Patients in both groups receive 8 mL/kg/hour of Ringer's lactate solution from 30 minutes prior to induction of anaesthesia through the end of surgery, when the rate will be decreased to 100 mL/hour. In addition, boluses of colloid will be given to different protocol group according to the study arm to which the patient allocated.Postoperative care and discharge criteria were predefined using the hospital care map and protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients scheduled for total hip replacement at this institution.
* 2. American Society of Anaesthesiologists (ASA) physical status of III or VI.
* 3. Two or more risk factors according to risk index of Lee .

Exclusion Criteria:

* 1. Age under 70years old
* 2. idiopathic coagulopathy: with warfarin or heparin
* 3. systemic or local infection
* 4. unable to cooperate
* 5. spinal trauma or severe low back pain history
* 6. patient refusal.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
length of postoperative hospital stay | 28 days
  days from end of surgery to hospital discharge.

SECONDARY OUTCOMES:
postoperative complications and mortality | 28 days
  1. Major complications: Infection , Major cardiovascular complications , Pulmonary Embolism, Renal Failure, Anaemia requiring blood transfusion in the presence of shock.
  2. Minor complications: Hypotension (systolic blood pressure < 90 mmHg) requiring fluid boluses, Uncomplicated infections (not requiring intra-venous antibiotic therapy and with no signs of sepsis, i.e. uncomplicated urinary tract infections), Anemia requiring blood transfusions in the absence of shock.
  3. PONV: Postoperative Nausea and Vomiting
  4. delirium and postoperative cognitive dysfunction
  5. mortality

OTHER OUTCOMES:
information of hemodynamic and ScvO2 ,types and volumes of all fluids administered | 24 hours after operation

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD, PHD, Principal Investigator — Guangzhou First Municipal People's Hospital,Guangzhou Medical College
Locations (1):
- Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Gan TJ, Soppitt A, Maroof M, el-Moalem H, Robertson KM, Moretti E, Dwane P, Glass PS. Goal-directed intraoperative fluid administration reduces length of hospital stay after major surgery. Anesthesiology. 2002 Oct;97(4):820-6. doi: 10.1097/00000542-200210000-00012. PMID 12357146
- [Background] Mayer J, Boldt J, Wolf MW, Lang J, Suttner S. Cardiac output derived from arterial pressure waveform analysis in patients undergoing cardiac surgery: validity of a second generation device. Anesth Analg. 2008 Mar;106(3):867-72, table of contents. doi: 10.1213/ane.0b013e318161964d. PMID 18292432 (Retraction: PMID 21451067 Anesth Analg. 2011 May;112(5):1074)
- [Background] Cecconi M, Fasano N, Langiano N, Divella M, Costa MG, Rhodes A, Della Rocca G. Goal-directed haemodynamic therapy during elective total hip arthroplasty under regional anaesthesia. Crit Care. 2011;15(3):R132. doi: 10.1186/cc10246. Epub 2011 May 30. PMID 21624138
- [Background] Lees N, Hamilton M, Rhodes A. Clinical review: Goal-directed therapy in high risk surgical patients. Crit Care. 2009;13(5):231. doi: 10.1186/cc8039. Epub 2009 Oct 26. PMID 19863764
- [Background] Moore JM. Continuous spinal anesthesia. Am J Ther. 2009 Jul-Aug;16(4):289-94. doi: 10.1097/MJT.0b013e3181729d2a. PMID 19546804